CLINICAL TRIAL: NCT03274921
Title: Identification of BIOmarkers for Detection and Understanding of Cardiovascular Complications in Chronic Kidney Disease
Brief Title: Biomarkers of Cardiovascular Complications in Chronic Kidney Disease
Acronym: BioClaCK
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/16/8250; University Hospital Toulouse (Other Grant/Funding Number: Local grant)
Record Dates: First submitted 2017-09-01; First posted 2017-09-07 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Chronic Renal Disease
Keywords: cardiovascular complications; biomarkers
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiovascular complication: patients with history of CV complications in the past 4 years had biological determination
  Interventions: Diagnostic Test: Biological determination
- No cardiovascular complication: patients free of any CV complications had biological determination
  Interventions: Diagnostic Test: Biological determination

INTERVENTIONS:
Diagnostic Test: Biological determination — Evaluation of plasma accumulation of the 10 retention solutes with CV complications in CKD patients

SUMMARY:
Identification of new retention solutes associated with cardiovascular (CV) toxicity in Chronic Kidney Disease (CKD) patients will help to better understand the pathophysiological mechanisms at stake and to prevent CKD-associated mortality and morbidity. For a molecule to be defined as a toxic retention solute, plasma accumulation in the course of CKD has to be demonstrated but also proof needs to be made that plasma accumulation during CKD is indeed associated with an increased risk of CV complications. Moreover, precise determination of the plasma concentration has to be performed in order to later study in vitro and in vivo the toxic mechanisms involved. Based on previous results of plasma proteome analysis using mass spectrometry, a previous study has selected 10 promising protein candidates. These proteins accumulated in the plasma of patients during CKD progression and are known to be associated with CV events in non-CKD patients. The objective of the present study is now to 1) evaluate the association of the plasma accumulation of the 10 retention solutes with CV complications in CKD patients and 2) determine their plasma concentration using ELISA. One hundred and seventy six patients with advanced CKD will be included and divided in 2 groups: 44 patients with history of CV complications in the past 4 years and 132 patients free of any CV complications.

ELIGIBILITY:
Inclusion Criteria:

* patient with stage 4 or 5 CKD.

Exclusion Criteria:

* patient with stage 1, 2 or 3 CKD
* patient with solid tumor
* patient with malignant blood disease
* patient with acute kidney disease in the past 3 months
* patient with acute glomerulonephritis in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of patients consulting in University Hospital toulouse
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Plasma accumulation of new retention solutes | Day 0
  evaluate the plasma accumulation of the 10 retention solutes using mass spectrometry

SECONDARY OUTCOMES:
determine their plasma concentration | Day 0
  determine their plasma concentration using ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas FAGUER, MD, Principal Investigator — University Hosptial Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No